CLINICAL TRIAL: NCT01223833
Title: A Prospective Assessment of Loss of Grip Strength by Baseline BMI in Breast Cancer Patients Receiving Adjuvant Third-generation Aromatase Inhibitors and Tamoxifen
Brief Title: A Prospective Assessment of Loss of Grip Strength by Baseline BMI in Breast Cancer Patients Receiving Adjuvant Aromatase Inhibitors and Tamoxifen
Acronym: LOGRIBMET
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S51575
Record Dates: First submitted 2010-10-14; First posted 2010-10-19 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2010-11

CONDITIONS: Breast Cancer; Arthralgia
Keywords: breast cancer; postmenopausal; aromatase inhibitors; tamoxifen; arthralgia; IGF-I; BMI; grip strength
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- tamoxifen: 100 postmenopausal women with early breast cancer treated with tamoxifen in the adjuvant setting
- aromatase inhibitors: 200 postmenopausal women with early breast cancer treated with an aromatase inhibitor in the adjuvant setting

SUMMARY:
The Logribmet study is a prospective study that evaluate grip strength changes in both hands of postmenopausal women with breast cancer receiving treatment with tamoxifen or an aromatase inhibitor. Patients included in the study will undergo a grip strength measurement and receive a rheumatological questionnaire prior to the start of treatment, then at 3 and 6 months and at year 1 into therapy. Furthermore, BMI will be measured to assess if BMI is a predictor for the decrease in grip strength.

IGF-I, GH and IGFBP-3 serum levels will also be measured at all time points.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with early breast cancer who are scheduled to receive endocrine therapy with tamoxifen or any of the third-generation aromatase inhibitors, anastrozole, letrozole or exemestane.
2. No major rheumatological disorders such as severe rheumatoid arthritis.
3. Patients must have provided informed consent for participation in this study.

Exclusion Criteria:

1. Concomitant endocrine therapy for breast cancer.
2. Concomitant intake of sex hormone containing drugs such as hormone replacement therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal early breast cancer patients scheduled to start adjuvant hormonal therapy with any of the third generation aromatase inhibitors or tamoxifen in University Hospitals Leuven.
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2009-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To assess the effect of BMI on loss of grip strength measured by a modified sphygmomanometer with baseline, month 3, month 6 and month 12 measurements. | 1 year
  measurements occur at baseline, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
IGF-I, GH and IGFBP-3 levels | 1 year
  Serum levels of IGF-I, GH and IGFBP-3 will be measured at baseline, 3, 6 and 12 months after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neven, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium